CLINICAL TRIAL: NCT03799562
Title: Neurosteroid Intervention for PTSD in Iraq/Afghanistan-era Veterans
Brief Title: Neurosteroids for PTSD in Veterans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-004-18S; I01CX001784-01 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Depression; Pain; Clinical Trial; Veteran; Supplement
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Pain | interventions — Pregnenolone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the active study medication (pregnenolone) or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, double-blind, placebo-controlled trial. All roles will be masked with the exception of the research pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pregnenolone (Experimental): Placebo lead in 14 DAYS, followed by Pregnenolone 50 mg BID x 14 DAYS, followed by Pregnenolone 150 mg BID x 14 DAYS, followed by Pregnenolone 250 mg BID x thereafter for the remainder of the 8-week trial
  Interventions: Drug: Pregnenolone
- Placebo (Placebo Comparator): Same as pregnenolone (active study medication), except placebo dispensed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Pregnenolone 50 mg BID x 14 DAYS, followed by Pregnenolone 150 mg BID x 14 DAYS, followed by Pregnenolone 250 mg BID x thereafter for the remainder of the 8-week trial. Placebo will be identical to the pregnenolone arm, except placebo will be dispensed.
  Arms: Pregnenolone
Drug: Placebo — Same as pregnenolone (active study medication), except placebo dispensed.
  Arms: Placebo

SUMMARY:
This study seeks to determine if pregnenolone can improve symptoms of PTSD and other symptoms that commonly occur with PTSD in Iraq/Afghanistan-era Veterans. The total study duration is 10 weeks. Eligible Veterans with PTSD will receive either pregnenolone or placebo throughout the study duration and will complete mental and physical health assessments at each study visit. Eligible participants will attend 6 in-person study visits and receive several short "check-in" phone calls.

DETAILED DESCRIPTION:
BACKGROUND: There is an acute and urgent need to develop new and effective posttraumatic stress disorder (PTSD) pharmacotherapies, as there are currently only two FDA-approved medications for the treatment of PTSD (both of which are from the same drug class and have shown only moderate effect sizes in FDA registration trials). Many Veterans with PTSD thus remain symptomatic despite the availability of these treatments, increasing the likelihood of receiving pharmacological treatment interventions for which there is little or no empirical evidence. Multiple national and VA working groups focusing on PTSD have identified the critical need to address the paucity of PTSD pharmacotherapies, and have strongly recommended more randomized clinical trials to evaluate possible effective pharmacological treatments. Both preclinical and clinical data suggest that reductions in neurosteroids are involved in the pathophysiology of PTSD, and that ameliorating these deficits could potentially be clinically therapeutic - the proposed investigation targeting a neurosteroid intervention for the treatment of PTSD could thus be a promising research avenue. The investigators therefore propose to conduct a randomized clinical trial (RCT) to determine the efficacy of a neurosteroid intervention (pregnenolone) for PTSD and commonly co-occurring disorders in Iraq/Afghanistan-era Veterans, an understudied cohort that may be less treatment-refractory.

METHODS: This study will be a 10-week randomized, placebo-controlled, double-blind clinical trial of pregnenolone or matching placebo in Veterans with PTSD. The trial will include a 2-week single-blind placebo lead-in phase followed by 8 weeks of study medication (placebo or pregnenolone). Forty-five subjects meeting DSM-5 criteria for PTSD (as measured by a CAPS-5 score of 30) will be randomized to receive pregnenolone, and 45 subjects meeting DSM-5 criteria for PTSD will be randomized to receive placebo. The primary outcome for this RCT will be changes in total CAPS-5 score at Visit 6 for this modified intent-to-treat sample. Secondary clinical outcomes for this RCT include changes in pain intensity and functional interference, as measured by the Brief Pain Inventory, Short Form (BPI-SF) and depression symptoms by the Hamilton-Depression Rating Scale (HAM-D). Blood samples will be collected for serum analysis at all study visits and frozen in a -80 degree freezer. Upon completion of the study, samples will be thawed and analyzed using Gas Chromatography/Mass Spectrometry for neurosteroid analyses and inflammatory markers will be quantified. Genetic analyses will be conducted to determine therapeutic response.

PREDICTED RESULTS: The investigators hypothesize that treatment with pregnenolone will be efficacious in Iraq/Afghanistan-era Veterans with PTSD, and will significantly reduce PTSD symptoms as assessed by the CAPS-5 (primary endpoint) compared to placebo. Secondary endpoints will include the assessment of conditions that frequently co-occur with PTSD; specifically, the investigators hypothesize that pregnenolone will also demonstrate efficacy for co-occurring chronic pain symptoms and depression symptoms. The investigators hypothesize that increases in pregnenolone and other neurosteroids (and decreases in inflammatory markers) will predict improvements in PTSD, depression, and chronic pain symptoms. The investigators also hypothesize that neurosteroids are dysregulated in PTSD, and that specific SNPs of genes coding for neurosteroidogenic enzymes will be associated with therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of PTSD with CAPS-5 Total Score 3
* Females will be required to use a medically and study approved contraceptive or otherwise not be of child-bearing potential

  * Birth control methods must be non-hormonal
* No anticipated need to alter psychiatric medications for duration of study involvement
* Ability to participate fully in the informed consent process

Exclusion Criteria:

* History of allergy to pregnenolone
* Medical disorders that may preclude safe administration of pregnenolone or exacerbate PTSD symptoms
* Current suicidal or homicidal ideation necessitating clinical intervention or representing an imminent concern

  * Prior suicide attempt history or suicidal ideation that does not require clinical intervention or represent an imminent concern is permitted
* Serious unstable medical illness, such as:

  * history of cerebrovascular accident
  * prostate
  * uterine or breast cancer
  * others (at the discretion of the PI and medical oversight team)
* Medical conditions not well controlled will be excluded, at the discretion of the PI and Medical Team
* Standard pharmacological interventions for PTSD will not be exclusionary, including, but not limited to:

  * antidepressant medications such as SSRIs, SNRIs, tricyclics, bupropion, mirtazapine, venlafaxine, and nefazodone
  * mood stabilizers such as carbamazepine, divalproex, lamotrigine, topiramate
  * atypical antipsychotics, and other agents including prazosin
  * However, there may be no changes in psychotropic medications for PTSD 4 weeks prior to study randomization
* Benzodiazepine use
* Current diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition other than mild TBI (assessed at screening)
* Initiation or change in psychotherapy within 3 months of randomization

  * i.e., psychotherapy must be stable for 3 months prior to study start
* Participants on hormonal therapies such as finasteride or hormonal birth control
* Female participants who are pregnant or breast-feeding
* As indicated by the DSM-5, moderate or severe Substance Use Disorders (excluding caffeine and tobacco) within 1 month of study entry

  * Mild Alcohol Use Disorder is not exclusionary, at the judgment of the PI and her medical team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale for DSM-5 (Visit 6-Baseline) | Through study completion, an average of 5 years
  The CAPS is the gold standard in PTSD assessment. The CAPS-5 is a 30-item structured interview that can be used to make a diagnosis of PTSD and assess PTSD symptoms. It assesses the intensity and frequency of PTSD symptoms. Scores range from 0-80; higher score indicates greater severity.

SECONDARY OUTCOMES:
Change in Brief Pain Inventory, Short Form (Visit 6-Baseline) | Through study completion, an average of 5 years
  The Brief Pain Inventory, Short Form (BPI-SF) is a self-reported scale that measures the severity of pain and the interference of pain on function. The scores range from 0 (no pain) to 10 (pain as severe as you can imagine). There are 4 questions assessing worst pain, least pain, average pain in the past 24 hours, and the pain right now. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
Change in Hamilton-Depression Inventory (Visit 6-Baseline) | Through study completion, an average of 5 years
  The HAM-D measures the severity of depressive symptoms. It is a checklist of 17 items that are ranked on a scale of 0-4 or 0-2. The range for the total score (which is the sum of the scores of all 17 items) is 0-52; a higher score indicates greater severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Naylor, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03799562/ICF_000.pdf